CLINICAL TRIAL: NCT04223401
Title: Personalized Trimodal Prehabilitation for Gastrectomy
Brief Title: Prehabilitation for Gastrectomy
Acronym: PREFOG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other)
Collaborators: Vilnius University (Other); Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): Patients in the experimental group will undergo prehabilitation before the elective surgery for gastric cancer.
  Interventions: Other: Prehabilitation
- Control group (No Intervention): Patients in the control group will not undergo prehabilitation.

INTERVENTIONS:
Other: Prehabilitation — Patients will undergo 6 Minutes Walking Test (6-MWT), spiroergometry (VO2 max; AT), a grip strength test, a timed Up & Go (TUG) test, 10 m sprint test and sit to stand test before and after prehabilitation. The trimodal intervention will involve:
  1. Nutritional intervention
  2. Psychological intervention
  3. Exercise intervention
  Arms: Prehabilitation group

SUMMARY:
Prehabilitation has been demonstrated to be an effective strategy to improve outcomes in patients undergoing some of the abdominal operations. It may increase the physical capacity of the patient, improve postoperative quality of life and even decrease the postoperative morbidity. Currently, the most effective strategy seems to be a trimodal prehabilitation which includes: 1) Nutritional support 2) Psychological support and 3) Physical training.

DETAILED DESCRIPTION:
This study will investigate personalized trimodal prehabilitation for patients undergoing gastrectomy for gastric cancer.

Prehabilitation group:

Patients will undergo 6 Minutes Walking Test (6-MWT), spiroergometry (VO2 max; AT), a grip strength test, a timed Up & Go (TUG) test, 10 m sprint test and sit to stand test before and after prehabilitation. The trimodal intervention will involve:

1. Nutritional intervention: The dietetic physician will perform physical examination and evaluation of the nutritional status to provide individualized care to each patient. Patients will receive personalized recommendations for the prevention or correction of malnutrition.
2. Psychological intervention: Patients will undergo consultation by specialized onco-psychologist. The anxiety and depression level will be evaluated by HAD score and patients will be trained to perform techniques, such as relaxation to reduce and manage anxiety on at home basis.

   The psychologist also will enhance patients' motivation to comply with the exercise and nutritional aspects of the intervention.
3. Exercise intervention: Patients will be consulted by PM&R physicians and physiotherapists and personalized exercise plans will be developed according to the results of 6MWT, AT and VO2peak. Exercises will focus on skeletal muscles and cardiopulmonary function training and the exercises feasible at home basis will be selected. All patients will undergo three supervised training sessions to learn the correct exercise techniques.

All patients will be routinely contacted to ensure compliance with prehabilitation program.

Patients scheduled for surgery first by multidisciplinary tumor board will undergo 4 weeks prehabilitation program, while patients scheduled for perioperative chemotherapy will undergo prehabilitation while neoadjuvant treatment will be administered.

Control group:

Patients will also undergo 6 Minutes Walking Test (6-MWT), spiroergometry (VO2 max; AT), a grip strength test, a timed Up & Go (TUG) test, 10 m sprint test and sit to stand test before surgery or before and after neoadjuvant chemotherapy. Patients will not undergo prehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient agrees to participate in a clinical study
* Patient requires surgical treatment for gastric cancer

Exclusion Criteria:

* Patient requiring surgical treatment for recurrent gastric cancer
* Patient condition not allowing to postpone surgery for at least 4 weeks
* Patients physical or mental condition which will not allow the patient to participate in prehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative morbidity rate by Clavien-Dindo | At 90 days postoperatively

SECONDARY OUTCOMES:
Physical status by Spiroergometry | Baseline, pre-surgery, 3, 6 and 12 months after surgery
Physical status by International Physical Activity Questionnaire (IPAQ) | Baseline, pre-surgery, 3, 6 and 12 months after surgery
Postoperative mortality rate | At 30 and 90 days postoperatively
Nutritional status by albumin level | Baseline, pre-surgery, 3, 6 and 12 months after surgery
Quality of Life by EORTC questionnaires | Baseline, pre-surgery, 3, 6 and 12 months after surgery
Percentage of patients reaching the complete oncological treatment fixed in a multidisciplinary tumour board (including preoperative chemotherapy, surgery and postoperative chemotherapy) | 12 months after surgery
Physical status by grip strength test | Baseline, pre-surgery, 3, 6 and 12 months after surgery
Physical status by 6 minutes walk test | Baseline, pre-surgery, 3, 6 and 12 months after surgery
Physical status by the sit to stand test | Baseline, pre-surgery, 3, 6 and 12 months after surgery
Physical status by the timed up&go test | Baseline, pre-surgery, 3, 6 and 12 months after surgery
Psychological status by Hospital Anxiety and Depression Scale (HADS). | Baseline, pre-surgery, 3, 6 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kestutis Strupas, MD PhD Prof., Principal Investigator — Vilnius University
Locations (2):
- Lithuania (2):
  - National Cancer Institute, Vilnius
  - Vilnius University hospital Santaros klinikos, Vilnius

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bausys A, Luksta M, Anglickiene G, Maneikiene VV, Kryzauskas M, Rybakovas A, Dulskas A, Kuliavas J, Stratilatovas E, Macijauskiene L, Simbelyte T, Celutkiene J, Jamontaite IE, Cirtautas A, Lenickiene S, Petrauskiene D, Cikanaviciute E, Gaveliene E, Klimaviciute G, Rauduvyte K, Bausys R, Strupas K. Effect of home-based prehabilitation on postoperative complications after surgery for gastric cancer: randomized clinical trial. Br J Surg. 2023 Nov 9;110(12):1800-1807. doi: 10.1093/bjs/znad312. PMID 37750588
- [Derived] Bausys A, Luksta M, Kuliavas J, Anglickiene G, Maneikiene V, Gedvilaite L, Celutkiene J, Jamontaite I, Cirtautas A, Lenickiene S, Vaitkeviciute D, Gaveliene E, Klimaviciute G, Bausys R, Strupas K. Personalized trimodal prehabilitation for gastrectomy. Medicine (Baltimore). 2020 Jul 2;99(27):e20687. doi: 10.1097/MD.0000000000020687. PMID 32629639